CLINICAL TRIAL: NCT06286397
Title: Topical Anti-Androgens in Pilonidal Sinus Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 855173
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pilonidal Disease; Pilonidal Disease of Natal Cleft; Pilonidal Sinus; Pilonidal Cyst
Keywords: Pilonidal Cyst; Pilonidal Sinus; Clascoterone; Androgen
MeSH Terms: conditions — Pilonidal Sinus | interventions — Clascoterone

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clascoterone Treatment (Experimental): Participants will apply 1% clasocterone cream to the affected area twice daily got a total of 12 weeks with assessment visits at weeks 0, 4, 8, and 12. At assessment visits participants will have medical photography of the diseased area, be administered a dermatology-specific quality of life questionnaire, and be assessed for any side effects.
  Interventions: Drug: 1% Clascoterone
- Placebo Treatment (Placebo Comparator): Participants will apply a vehicle cream matched in texture, appearance, and odor to clacoterone to the affected area twice daily got a total of 12 weeks with assessment visits at weeks 0, 4, 8, and 12. At assessment visits participants will have medical photography of the diseased area, be administered a dermatology-specific quality of life questionnaire, and be assessed for any side effects.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: 1% Clascoterone — Application of 1% clascoterone cream twice daily to affected area for 12 weeks.
  Arms: Clascoterone Treatment
Drug: Vehicle Cream — Application of a vehicle cream to the natal cleft twice daily for 12 weeks
  Arms: Placebo Treatment

SUMMARY:
The goal of this randomized clinical trial is to test the topical drug clascoterone in patients with pilonidal disease, which is a common, benign skin condition of the gluteal cleft. The main questions it aims to answer are:

* Does clascoterone improve the severity of pilonidal disease as scored by a physician?
* Does clascoterone improve patient symptoms due to pilonidal disease?
* Does clascoterone improve the inflammation seen under the microscope in pilonidal disease removed at surgery Participants will apply clascoterone or a placebo cream to the diseased area for 3 months. They will be assessed every 4 weeks for disease severity assessed by a physician viewing patient photos and a symptom-based survey.

Researchers will compare participants who received clascoterone treatment to those who received placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blinded placebo-controlled trial. Recruitment The investigators will recruit patients from the University of Pennsylvania colorectal surgery clinics which consist of six high-volume surgeons and five advance practice providers across three hospitals serving a major metropolitan area. Patients considered for elective surgery will be recruited for the study and undergo a thorough informed consent process. Patients with asymptomatic disease and those with acute abscesses will be excluded as will patients who are pregnant or concurrently on a systemic anti-androgen (i.e. spironolactone). At the intake visit, patients will undergo a 1:1 randomization performed by the University of Pennsylvania's Investigational Drug Service (IDS). Recruited subjects will receive clascoterone or a vehicle cream matched for consistency, color, and container so that both subject and investigator are blinded to the assignment. At the intake visit, subjects will be advised to apply cream to cover the affected area twice daily for 12 weeks. At the intake visit, baseline disease assessment will be obtained including demographics, height and weight, medication usage, and personal history of PSD such as disease onset and prior procedures. Baseline disease measurements and medical photography will be obtained. Photographs will be taken with a dedicated camera, patients given a codified study ID, and data entered into a deidentified, HIPAA- compliant database.

I. Objective assessment of Disease Severity: Medical photography and analysis To objectively evaluate PSD, the investigators will obtain physical measurements of disease extent (left to right, cranial to caudal) and obtain disease photographs at baseline and weeks 4, 8, and 12. Photographs will be collected, deidentified, and provided to two colorectal surgeons for scoring. Surgeons will be asked to compare each timepoint to baseline and rate the PSD severity as significantly worsened, mildly worsened, unchanged, mildly improved, or significantly improved. Discrepant evaluations between surgeons will be referred to a third blinded surgeon.

II. Assessment of Dermatology Quality of Life Randomized subjects will be administered the Dermatology Life Quality Index (DLQI) at baseline and at 4, 8, and 12 weeks. The DLQI is a 10-question survey scored from 0-30 that has been applied widely across multiple dermatologic conditions and covers a range of potential quality of life impacts over a weekly basis. Specifically, the DLQI inquires about the impact of skin disease on symptoms ("Over the past week, how itchy, painful, or stinging has your skin been?"), daily activities, leisure, work and school, and personal relationships, as well as a question of impact of treatment ("Over the last week, how much of a problem has the treatment of your skin been?"). Subjects respond Very much, A lot, A little, or Not at all for descending scores of 3 to zero. A score at or above 10 is considered a significant impact on quality of life. Responses to the individual questions will be summed and responses compared between groups after unblinding at data analysis.

III. The investigators anticipate that a large portion of subjects in both groups will ultimately undergo surgery. Those that undergo surgery within 4 weeks will be selected for these analyses, on the hypothesis that the effect of clascoterone may subside at a longer interval. At surgery, blinded investigators will measure the left-right, cranial-caudal, and superficial-deep measurements of the excisional defect with a sterile ruler. The investigators will then follow patients with chart review in the electronic medical record for 8 weeks postoperatively to assess for immediate wound complications such as cellulitis, wound separation, abscess, and early recurrence.

III. Assessment of Cutaneous Inflammation A full thickness representative sample of the excised pilonidal cyst and adjacent normal tissue will be obtained at operation, fixed in formalin and delivered to the skin phenomics core of the University of Pennsylvania Skin Biology Disease Research Core (SBDRC). Following de-paraffination, rehydration, antigen retrieval, and blocking as necessary, SBDRC-validated antibodies will be applied to characterize the inflammatory infiltrate, specifically anti- CD3 (T- cells and Natural Killer Cells), anti-CD4 (helper T-cells), anti-CD8 (cytotoxic T-cells), anti-CD68 (macrophages), anti-CD79 (B cells). Investigators blinded to treatment groups will assess the specimens for epidermal, dermal, and subcuticular inflammatory infiltrates, hyperkeratosis, and follicular hyperplasia. Antibody-positive cells will be counted in six randomly selected fields under a light microscope at 400x magnification. Cell counts will be tallied and means and standard deviations compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Diagnosis of Pilonidal Disease
* Willingness to comply with study procedures and availability for duration of study
* Ability to apply topical medications and willing to adhere to regimen

Exclusion Criteria:

* Current use of any topical medication to natal cleft
* Presence of pilonidal-associated abscess
* Pregnancy or lactation
* Allergic reaction to components of 1% clascoterone cream
* Febrile illness within 7 days
* Treatment with another investigational drug within three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Physician-Assessed Disease Severity Assessment | From enrollment to the end of treatment at 12 weeks
  To objectively evaluate PSD, the investigators will obtain physical measurements of disease extent (left to right, cranial to caudal) and obtain disease photographs at baseline and weeks 4, 8, and 12. Photographs will be collected, deidentified, and provided to two colorectal surgeons for scoring. Surgeons will be asked to compare each timepoint to baseline and rate the PSD severity as significantly worsened, mildly worsened, unchanged, mildly improved, or significantly improved. Discrepant evaluations between surgeons will be referred to a third blinded surgeon. Data will be collated and analyzed in two fashions: as a 6-point ordinal outcome and collapsed into a dichotomous outcome with severely worsened to no change as a negative outcome and improvement as a positive outcome.
Dermatology Life Quality Index | From enrollment to the conclusion of treatment at 12 weeks
  Randomized subjects will be administered the Dermatology Life Quality Index (DLQI) at baseline and at 4, 8, and 12 weeks. The DLQI is a 10-question survey scored from 0-30 that has been applied widely across multiple dermatologic conditions and covers a range of potential quality of life impacts over a weekly basis. Specifically, the DLQI inquires about the impact of skin disease on symptoms (Example: "Over the past week, how itchy, painful, or stinging has your skin been?"), daily activities, leisure, work and school, and personal relationships, as well as a question of impact of treatment ("Over the last week, how much of a problem has the treatment of your skin been?"). Subjects respond Very much, A lot, A little, or Not at all for descending scores of 3 to zero. A score at or above 10 is considered a significant impact on quality of life.

SECONDARY OUTCOMES:
Subcutaneous Inflammation | From 12 weeks to 16 weeks after enrollment, only in patients who undergo surgery
  The investigators anticipate that a large portion of subjects will ultimately undergo surgery. Those that undergo surgery within 4 weeks will be selected. At surgery, blinded investigators will measure the excisional defect. The investigators will then follow patients with chart review in the electronic medical record for 8 weeks postoperatively to assess for immediate wound complications. A full thickness representative sample of the excised pilonidal cyst will analyzed including: antibodies against CD3, CD4, CD8, CD68, and D79. Investigators will assess the specimens for hyperkeratosis, and follicular hyperplasia.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hebert A, Thiboutot D, Stein Gold L, Cartwright M, Gerloni M, Fragasso E, Mazzetti A. Efficacy and Safety of Topical Clascoterone Cream, 1%, for Treatment in Patients With Facial Acne: Two Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2020 Jun 1;156(6):621-630. doi: 10.1001/jamadermatol.2020.0465. PMID 32320027
- [Background] Kalabalik-Hoganson J, Frey KM, Ozdener-Poyraz AE, Slugocki M. Clascoterone: A Novel Topical Androgen Receptor Inhibitor for the Treatment of Acne. Ann Pharmacother. 2021 Oct;55(10):1290-1296. doi: 10.1177/1060028021992053. Epub 2021 Feb 3. PMID 33533262
- [Background] Hargis A, Yaghi M, Maskan Bermudez N, Lev-Tov H. Clascoterone in the treatment of mild hidradenitis suppurativa. J Am Acad Dermatol. 2024 Jan;90(1):142-144. doi: 10.1016/j.jaad.2023.08.064. Epub 2023 Sep 2. No abstract available. PMID 37660976